CLINICAL TRIAL: NCT00681785
Title: Thromboseprophylaxe Mit Niedermolekularem Heparin Bei Transurethralen Eingriffen
Brief Title: Thrombophylaxis in Transurethral Surgery With Dalteparine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Maurer Patrick, Dr, Department of Urology, Kantonsspital Liestal
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 269/05
Record Dates: First submitted 2008-04-21; First posted 2008-05-21 (Estimated); Last update posted 2008-05-21 (Estimated); Status verified 2008-05

CONDITIONS: Thrombophylaxis in Transurethral Surgery
Keywords: thrombophylaxis and transurethral surgery
MeSH Terms: interventions — Dalteparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): 5000IE dalteparine
  Interventions: Drug: dalteparine (Fragmin)
- B (Placebo Comparator): NaCL 0.9%
  Interventions: Drug: dalteparine (Fragmin)

INTERVENTIONS:
Drug: dalteparine (Fragmin) — transurethrals surgery with and without dalteparine
  Other Names: Dlateparine=Fragmin

SUMMARY:
The rationale for thrombophrophylaxis is well known. Without prophylaxis the incidence of objectivlely confirmed, hospital-acquired deep venous thrombosis is approximately 10% to 40% among medical or general surgical patients. In urology the prevalence is 15-40%. The Seventh ACCP Conference on Antithrombotic and Thrombolytic Therapy1 recommend against specific prophylaxis in patients undergoing transurethral procedures. Our study is the first double-blind, placebo-controlled study with Dalteparine as thrombophrophylaxis in transurethral surgery. The aim of the study is to proof that thrombophrophylaxis causes not more complications in transurethral surgery than without.

DETAILED DESCRIPTION:
The aim of our study is to proof that transurethral surgery under thrombophylaxis with dalteparine is safe. The study design is double-blind placebo controlled.

ELIGIBILITY:
Inclusion Criteria:

* transurethral surgery

Exclusion Criteria:

* oral anticoagulation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2006-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Blood loss | intraoperativ, 6 hours post op and 3 days postop

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Gasser, Prof, Study Chair — Department of Urology Liestal
Locations (1):
- Urologische Universitätsklinik beider Basel, Liestal, Switzerland